CLINICAL TRIAL: NCT00475930
Title: Chlorhexidine Impregnated Cloths to Prevent Skin and Soft Tissue Infections in Marine Officer Candidates: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Chlorhexidine Impregnated Cloths to Prevent Skin and Soft Tissue Infections in Marine Officer Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HU87F7
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Staphylococcus Aureus; Community-acquired Infections; Staphylococcal Skin Infections
Keywords: MRSA; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections; Community-Acquired Infections; Staphylococcal Skin Infections | interventions — chlorhexidine gluconate; Chromogranins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 2% chlorhexidine gluconate impregnated cloths, self applied three times weekly
  Interventions: Drug: 2% chlorhexidine gluconate (CHG) impregnated cloths
- 2 (Placebo Comparator): Comfort Bath cloths, self applied three times weekly
  Interventions: Drug: Comfort Bath cloths (placebo cloths)

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate (CHG) impregnated cloths — self applied three times per week
  Other Names: Sage Products Inc.
  Arms: 1
Drug: Comfort Bath cloths (placebo cloths) — self applied three times weekly
  Other Names: Sage Products Inc.
  Arms: 2

SUMMARY:
Outbreaks of skin and soft tissue infections (SSTI) related to community associated Methicillin-resistant Staphylococcus aureus (MRSA) have become increasingly common in military training units. Risk factors for MRSA related SSTI such as crowding, poor hygiene and shared equipment are often hard to avoid in a military training environment, often designed to simulate battlefield conditions.

It has recently been demonstrated that military recruits colonized with MRSA may be at increased risk of developing SSTI. Studies in the hospital environment have shown that decolonizing inpatients known to carry MRSA decreases the rates of MRSA related infections in the treated individuals and also in their inpatient unit as a whole.

The investigators propose a randomized, double blind, placebo controlled trial to:

1. Evaluate the effectiveness, feasibility, and safety of chlorhexidine body cloths, self-administered three times weekly, in preventing SSTI among recruits in military training facilities; and
2. Evaluate the effectiveness of chlorhexidine body cloths in decreasing rates of Staphylococcus aureus colonization among military recruits.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in US Marine Officer Candidates School
* Age 18-35 years
* Provide documented informed consent and HIPAA authorization

Exclusion Criteria:

* Is currently taking oral antibiotics and will continue to take antibiotics during the study (such as antibiotics used to treat acne)
* Has a known or suspected allergy or intolerance to chlorhexidine (Hibistat, Hibiclens)
* Is currently using certain skin products and is uninterested in stopping use of the products during the study
* Pregnant or breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1563 (Actual)
Dates: Start 2007-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The rate of skin and soft tissue infections among platoons enrolled in OCS. | May - Nov 2007

SECONDARY OUTCOMES:
The rate of new S. aureus colonization of the nares and axilla among platoons enrolled in OCS. | May- Nov 2007

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Whitman, DO, Principal Investigator — National Naval Medical Center
Locations (1):
- Officer Candidates School - Marine Corps Base Quantico, Quantico, Virginia, United States

REFERENCES:
- [Derived] Whitman TJ, Herlihy RK, Schlett CD, Murray PR, Grandits GA, Ganesan A, Brown M, Mancuso JD, Adams WB, Tribble DR. Chlorhexidine-impregnated cloths to prevent skin and soft-tissue infection in Marine recruits: a cluster-randomized, double-blind, controlled effectiveness trial. Infect Control Hosp Epidemiol. 2010 Dec;31(12):1207-15. doi: 10.1086/657136. Epub 2010 Oct 28. PMID 21028984